CLINICAL TRIAL: NCT06495242
Title: Outcome of Direct Pulp Capping Compared to Partial Pulpotomy in the Management of Carious Pulp Exposures in Mature Teeth: A Randomized Clinical Trial
Brief Title: Direct Pulp Capping Compared to Partial Pulpotomy in Carious Pulp Exposures
Acronym: Pulp cap
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Nessrin Taha, Professor, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131/2023
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Deep Caries
Keywords: Caries, pulpitis, direct pulp capping, partial pulpotomy,, pain
MeSH Terms: conditions — Pulpitis; Pain

STUDY DESIGN:
Intervention Model Description: Parallel randomized clinical trial including 2 treatment groups with 1;1 allocation ration
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the participants are blinded to the type of treatment provided, the care provider is masked only during the early stages of teh procedure but subsequently masking is not possible due to different treatment protocols.
  Block randomization. and sealed envelop technique are used. Principal investigator and evaluator are blinded to the type of treatment provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct pulp capping (Active Comparator): After caries excavation and pulp exposure, the cavity is disinfected . the capping material is applied and the tooth is restored.
  Interventions: Procedure: Direct pulp capping and partial pulpotomy
- Partial pulpotomy (Active Comparator): After caries excavation and pulp exposure, 2-3 mm of the exposed pulp are cut . The capping material is applied and the tooth is restored.
  Interventions: Procedure: Direct pulp capping and partial pulpotomy

INTERVENTIONS:
Procedure: Direct pulp capping and partial pulpotomy — Two types of vital pulp therapy procedures
  Other Names: Partial pulpotomy

SUMMARY:
This a prospective randomized clinical trial that compare vital pulp therapy procedures in permanent teeth with carious pulp exposure. Patients are recruited from the dental teaching clinics at JUST following preset inclusion criteria. They are subsequently randomly assigned to one of treatment procedures. Clinical and radiographic follow up is performed after 6 months and yearly up to 5 years.

DETAILED DESCRIPTION:
Background: Deep carious lesions are commonly encountered in both adults and children with no clear consensus on the ideal clinical management. Vital pulp therapy including direct pulp capping and pulpotomy is increasingly considered in the management of carious pulp exposures when the clinical diagnosis is reversible pulpitis with variable reports of success rates with different materials used and different diagnostic categories.

Aims: The aims of this study are to evaluate the clinical and radiographic outcomes of direct pulp capping and partial pulpotomy in deep carious lesions of mature permanent teeth using a calcium silicate based material (Biodentine, Septodont, France), and to investigate the relationship between matrix metalloproteinase (MMP 9) levels in the pulpal blood and the outcome of these procedures.

Methods: 120 mature molar teeth in 120 patients with deep carious lesions exposing the pulps on the radiograph and with symptoms of reversible pulpitis will be included in the study. The teeth will be subsequently randomly divided into 2 groups (n=60). One group will receive direct pulp capping and composite restoration, and the second group will receive partial pulpotomy and composite restoration. Pulpal blood will be collected from the exposure site and will be tested for the level of MMP9 using special ElISA kit. Preoperative and postoperative pain level at 48 hours and 7 days will be evaluated on a scale from 0-10.

The treated teeth will be further evaluated clinically and radiographically at 6 and 12 months follow up and yearly afterward. The relationship of the outcome to the level of MMP9 will be investigated. The results will be statistically analyzed using appropriate tests in the SPSS software.

Expected results: Since partial pulpotomy includes the removal of 2-3 mm of the exposed pulp tissue which is theoretically inflamed, it is expected to be more effective in alleviating the patient's symptoms and to have a higher success rate than simply pulp capping the carious exposure. High levels of MMP9 are also expected to have a correlation with the failure rate.

ELIGIBILITY:
Inclusion Criteria:

* Non -contributory medical history (ASA 1)
* Molar tooth with extremely deep caries extending>2/3 of dentin or exposing the pulp on the periapical radiograph
* The tooth should give positive response to cold testing
* Clinical diagnosis of reversible pulpitis with mild to moderate symptoms
* The tooth is restorable, probing pocket depth and mobility are within normal limits
* No signs of pulpal necrosis including sinus tract or swelling
* No radiographic evidence of periapical changes indicative of apical periodontitis

Exclusion Criteria:

Immature teeth

* Nonvital teeth
* Irreversible pulpitis and periapical periodontitis, i.e spontaneous and lingering pain.
* Inability to achieve hemostasis after 6 minutes of application of 5% NaOCl moist pellet
* No pulp exposure after nonselective caries removal

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Short term clinical outcome | one week
  Resolution of clinical symptoms

SECONDARY OUTCOMES:
long term outcome | 1-5 years
  Maintenance of pulp vitality

CONTACTS AND LOCATIONS:
Overall Officials: Prof Nessrin A Taha, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Faculty of Dentistry, Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Original data can be provided upon a reasonable request, and may be available after publication

REFERENCES:
- [Background] Taha NA, Albakri SW. Outcome and Prognostic Factors for Partial and Full Pulpotomy in the Management of Spontaneous Symptomatic Pulpitis in Carious Mature Permanent Teeth: A Randomized Clinical Trial. J Endod. 2024 Jul;50(7):889-898. doi: 10.1016/j.joen.2024.03.012. Epub 2024 Apr 5. PMID 38583758
- [Background] Taha NA, Khazali MA. Partial Pulpotomy in Mature Permanent Teeth with Clinical Signs Indicative of Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2017 Sep;43(9):1417-1421. doi: 10.1016/j.joen.2017.03.033. Epub 2017 Jun 30. PMID 28673494
- [Background] Taha NA, Al-Khatib H. 4-Year Follow-up of Full Pulpotomy in Symptomatic Mature Permanent Teeth with Carious Pulp Exposure Using a Stainproof Calcium Silicate-based Material. J Endod. 2022 Jan;48(1):87-95. doi: 10.1016/j.joen.2021.09.008. Epub 2021 Sep 24. PMID 34563506
- [Background] Taha NA, Al-Rawash MH, Imran ZA. Outcome of full pulpotomy in mature permanent molars using 3 calcium silicate-based materials: A parallel, double blind, randomized controlled trial. Int Endod J. 2022 May;55(5):416-429. doi: 10.1111/iej.13707. Epub 2022 Mar 17. PMID 35152464
- [Background] Taha NA, Ahmad MB, Ghanim A. Assessment of Mineral Trioxide Aggregate pulpotomy in mature permanent teeth with carious exposures. Int Endod J. 2017 Feb;50(2):117-125. doi: 10.1111/iej.12605. Epub 2016 Jan 30. PMID 26715408